CLINICAL TRIAL: NCT03824899
Title: The Application of UGT1A1 Genotype Combined With Pharmacokinetics of SN-38 in the Detection of Irinotecan-based Neoadjuvant Chemoradiotherapy in Patients With Advanced Rectal Cancer
Brief Title: UGT1A1 Combined With Pharmacokinetics of SN-38 in CPT-11-based CRT in Patients With Advanced Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-010
Record Dates: First submitted 2019-01-20; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: neoadjuvant chemoradiotherapy; irinotecan; SN-38

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT group (Experimental): Patients With Advanced Rectal Cancer receiving CPT-11-based CRT and blood concentration check
  Interventions: Diagnostic Test: Blood concentration check

INTERVENTIONS:
Diagnostic Test: Blood concentration check — Blood concentration check：the plasma concentration of SN-38 was detected by HPLC (high-performance liquid chromatography) at 1.5 h and 49.0 h after CPT-11 infusion

SUMMARY:
The study evaluates the associations between peak and valley concentrations of SN-38 with the efficacy and adverse effects of advanced rectal cancer patients carrying genotype (TA) 6 /(TA) 6 or (TA) 6 /(TA) 7 after neoadjuvant chemoradiotherapy with CPT-11.All participants will be scheduled to receive surgery 6-8 weeks after the completion of CRT. The primary end point are toxicity and pCR rate.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed adenocarcinoma
* clinical stage T3-4 and/or N+
* the distance from anal verge less than 12 cm
* without distance metastases
* performance status score: 0~1
* UGT1A1*28 6/6 or 6/7
* without previous anti-cancer therapy
* sign the inform consent

Exclusion Criteria:

* pregnancy or breast-feeding women
* serious medical illness
* baseline blood and biochemical indicators do not meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L, ALT/AST ≤2.5 ULN, Cr≤ 1 ULN
* DPD deficiency
* UGT1A1*28 7/7

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
the morbidity of hematological adverse events and diarrhea as assessed by CTCAE v4.0 | During the chemoradiation weekly，assessed up to 5 weeks
  the morbidity of hematological adverse events and diarrhea as assessed by CTCAE v4.0
pathological response rate | Surgery scheduled 6-8 weeks after the end of chemoradiation
  pathological complete response (pCR) was defined no viable cancer cell under the examination of surgical resection specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China